CLINICAL TRIAL: NCT00076414
Title: The Effect of Lopinavir/Ritonavir on Endothelial Function in Normal Volunteers
Brief Title: The Effect of Lopinavir/Ritonavir on Endothelial Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040085; 04-CC-0085
Record Dates: First submitted 2004-01-21; First posted 2004-01-22 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-09

CONDITIONS: Healthy
Keywords: Endothelial Function; Lopinavir/Ritonavir; HIV; Blood Flow Studies; Flow-Mediated Vasodilatation; Healthy Volunteer; HV
MeSH Terms: interventions — Acetylcholine; omega-N-Methylarginine

INTERVENTIONS:
Drug: Acetylcholine
Drug: L-NMMA

SUMMARY:
This study will examine how the anti-HIV protease inhibitor lopinavir/ritonavir (Kaletra® (Registered Trademark)) affects the function of the endothelium (lining of the arteries). Medications such as protease inhibitors can dramatically change the course of HIV infection in many patients; however, among their side effects is development of abnormal lipid levels resulting in high cholesterol and insulin resistance. These side effects may damage the lining of the arteries that supply blood to the heart, leading to premature coronary artery disease. The study will determine whether lopinavir/ritonavir directly affects endothelial function and whether it alters cholesterol levels, glucose tolerance, and markers of inflammation in people who take the drug for 4 weeks.

Healthy normal volunteers between 18 and 40 years of age may be eligible for this study. Candidates must be HIV-negative and have no history of heart disease, hypertension, or diabetes mellitus. They must not have smoked for at least 6 weeks before entering the study. Volunteers will be screened with a medical history, physical examination, blood tests (including a pregnancy test for women of childbearing potential), and electrocardiogram. In addition, candidates will have an oral glucose tolerance test (see description below).

Participants will undergo the following procedures:

* Lopinavir/ritonavir: 4 weeks (3 capsules twice a day) beginning study day 1
* Flow-mediated vasodilatation test (study days 0 and 29) - An ultrasound device for measuring the size of the brachial artery (artery in the upper arm) is placed just above the elbow. The size of the artery is measured before and 5 minutes after blood flow to the arm is stopped for 5 minutes, using a blood pressure cuff. The artery is also measured before and after taking nitroglycerin, a medicine that dilates blood vessels. These measurements tell how well the drug treatment works on the cells lining the brachial artery, which is an indicator of coronary artery function. This test takes about 1.5 hours.
* Forearm blood-flow test (study days 1 and 30): Small tubes are inserted into an artery and vein in the forearm at the inside of the elbow. Blood pressure cuffs are placed around the upper arm and wrist, and a strain gauge (a rubber band-like device) is placed around the forearm. When the blood pressure cuffs are inflated, blood flows into the forearm, stretching the strain gauge at a rate proportional to the blood flow. When the devices are in place, a salt water solution is injected in the small tube in the artery. After 20 minutes, small doses of the following drugs are given through the catheter at various intervals: 1) L-NMMA (blocks production of nitric oxide, a substance produced by the blood vessels that causes them to dilate); 2) sodium nitroprusside (dilates blood vessels, increasing blood flow); 3) acetylcholine (lowers blood pressure); and 4) acetylcholine plus L-NMMA. The effect of the different drugs on blood flow in the forearm is measured. The study takes about 2 hours to complete.
* Blood tests (screening and study days 1,15, 30, and 44)
* Electrocardiogram (at screening and on study day 30)
* Oral glucose tolerance test (at screening and on study day 30) - A blood sample is collected. Then, the subject drinks 300 milliliters of a glucose solution (a liquid that contains sugar dissolved in water). Two hours after drinking the solution, blood is drawn again to examine how the body responds to the increase blood sugar levels.

DETAILED DESCRIPTION:
With the advent of the highly active antiretroviral (ARV) therapy era, patients with human immunodeficiency virus (HIV) have had significantly decreased mortality and morbidity. Concomitant with more patients chronically taking antiretroviral therapy, there has been an increase in atherogenic lipoprotein profiles (high cholesterol, high triglycerides, low HDL's), insulin resistance, fat redistribution and coronary artery disease. HIV viral replication, anti-retroviral treatment regimens, lipids, glucose intolerance, host immune response or a combination of factors may contribute to the increase in cardiovascular risk factors. HIV positive patients, independent of the effect on lipids, appear to have increased cardiovascular risk. Studies are not entirely consistent, but the most convincing study to date, the D.A.D. study from EURO-SIDA, shows a 27% relative increased rate of myocardial infarction per year of exposure over the first seven years of ART.

Lopinavir-ritonavir is one of the most commonly used antiretroviral therapy. It also produces lipid abnormalities. Thus, an important part of the investigating factors contributing to atherosclerosis would be to determine if this drug can adversely influence endothelial cells in the absence of HIV infection or low CD4 counts. This would suggest that this drug directly or indirectly could predispose to atherosclerosis. Endothelial function is an important contributor to atherosclerosis. Invasive and non-invasive methods to evaluate endothelial cell function have been validated as predictors of coronary artery disease. These techniques have been used at NIH for clinical investigation for many years.

This protocol is designed to determine whether there is a pathologic effect on endothelial function from the lopinavir/ritonavir. By measuring endothelial function in HIV non-infected subjects both before and after four weeks of therapy, we will be able to investigate whether the medications have a direct toxic effect on the endothelium. Collection of metabolic data will allow us to evaluate whether endothelial function occurs in conjunction or separate from lipoprotein and glucose metabolic changes. As ARV options increase, it may be possible to choose specific regimens that may minimize acceleration of cardiovascular risk factors associated with endothelial dysfunction, especially in patients with other cardiovascular risk factors. These findings may help elucidate the pathophysiology of premature cardiovascular disease in HIV positive patients and also plan interventions to minimize endothelial dysfunction and subsequent cardiovascular disease.

ELIGIBILITY:
INCLUSION CRITERIA:

Age 18-40.

Healthy by medical history and physical examination.

Negative serum pregnancy test for females.

Females willing to use two forms of birth control including barrier contraception during period of study (lopinavir/ritonavir decreases ethinyl estradiol levels).

Able to provide informed consent.

Laboratory values on screening visit within: AST less than 40 units/liter, serum creatinine less than 1.5mg/dl; CPK less than 387, hemoglobin greater than 11.0 g/dL (females) or greater than 12.6 g/dL (males), platelets greater than 154,000/mm(3), total bilirubin less than or equal to 1.5 mg/d

Total cholesterol less than 200 mg/dL, LDL cholesterol less than 160 mg/dL, HDL cholesterol greater than 30mg/dL, triglycerides less than 200 mg/dL.

Non-smoker or not having smoked for the past 6 weeks.

Negative for HIV by ELISA within 4 weeks of study participation.

EXCLUSION CRITERIA:

Concomitant therapy with any prescription, over-the-counter or alternative medication except intermittent use of acetaminophen, non-steroidal anti-inflammatory medications, loperamide or oral contraceptives.

Inability to obtain venous access for sample collection.

Presence of diabetes mellitus or fasting blood sugar greater than 126 mg/dL, or abnormal oral glucose tolerance test (2 hour post blood sugar greater than 200 mg/dL).

Human immunodeficiency virus (HIV) infection.

Cardiac disease, congestive heart disease, coronary artery disease, angina, carotid stenosis, peripheral vascular disease, cerebrovascular disease, myocardial disease, clinically significant valvular heart disease.

Any other condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the investigator.

Hypertension (systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg) on screening visit.

Observed abnormalities on EKG tracings that are significant in the opinion of the investigator (examples include, AV block, multifocal atrial tachycardia, frequent premature ventricular contractions, etc.).

Hypotension (systolic blood pressure less than 80 mmHG).

Pregnant or breastfeeding female.

Inability to abstain from caffeine use (coffee, tea or soda) or alcohol for 12 hours prior to a blood flow study until the conclusion of the study.

Heavy alcohol ingestion (4 or more drinks a day) or current substance abuse.

Hypo or hyper thyroidism.

Allergy to lidocaine.

History of hepatitis or other liver disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-01; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Duong M, Buisson M, Cottin Y, Piroth L, Lhuillier I, Grappin M, Chavanet P, Wolff JE, Portier H. Coronary heart disease associated with the use of human immunodeficiency virus (HIV)-1 protease inhibitors: report of four cases and review. Clin Cardiol. 2001 Oct;24(10):690-4. doi: 10.1002/clc.4960241011. PMID 11594416
- [Background] Carr A, Samaras K, Thorisdottir A, Kaufmann GR, Chisholm DJ, Cooper DA. Diagnosis, prediction, and natural course of HIV-1 protease-inhibitor-associated lipodystrophy, hyperlipidaemia, and diabetes mellitus: a cohort study. Lancet. 1999 Jun 19;353(9170):2093-9. doi: 10.1016/S0140-6736(98)08468-2. PMID 10382692
- [Background] Stein JH, Klein MA, Bellehumeur JL, McBride PE, Wiebe DA, Otvos JD, Sosman JM. Use of human immunodeficiency virus-1 protease inhibitors is associated with atherogenic lipoprotein changes and endothelial dysfunction. Circulation. 2001 Jul 17;104(3):257-62. doi: 10.1161/01.cir.104.3.257. PMID 11457741